CLINICAL TRIAL: NCT04862364
Title: Turkish Validation of Endometriosis Health Profile -30 (EHP-30) Test
Brief Title: Turkish Validation Study of Endometriosis Health Profile -30 (EHP-30) Test
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Engin Oral (Unknown)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ehp-30turkishvalidation
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Endo Patients with Endometriosis Health Profile -30 (EHP-30) Test — The appointment of the patients consists of patients who were surgically diagnosed with Endometriosis in our clinic.

SUMMARY:
For the Turkish validation Study of the Endometriosis Health Profile test (EHP-30) consisting of 30 questions, this 30-question test will be applied to 228 patients after 2 different translations to be applied after the translation of this 30-question test sworn translator to the patients who have been surgically diagnosed with endometriosis.

DETAILED DESCRIPTION:
The appointment of the patients consists of patients who were surgically diagnosed with Endometriosis in our clinic. English and Turkish translation will be verified after 2 different sworn translators.

ELIGIBILITY:
Inclusion Criteria:

* being surgically diagnosed with endometriosis
* Age between 18- 45
* not being pregnant

Exclusion Criteria:

* have been diagnosed with endometriosis by ultrasound
* above 45 and under 18 years old
* use psichiatrig drugs
* being diagnosed with a psychiatric illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with Endometriosis(surgicallay diagnosed)
Study Population: Female patients between the ages of 18-45 who were surgically diagnosed with endometriosis in our clinic will be included in the study. Persons with a known psychiatric illness, pregnant or using anti-depressant medication will be excluded from the study. Patients will be asked the questions of the online EHP-30 form and the answers given will be evaluated in terms of validation.
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Turkish Validation of Endometriosis Health Profile -30 (EHP-30) Test | 3 months
  The Turkish validation study of the Endometriosis Health Profile -30EHP-30 test, which shows the general quality of life of endometriosis patients, will be performed and the use of Turkish language will be provided.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided